CLINICAL TRIAL: NCT06277934
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled Study of RGT001-075 Compared With Placebo in Adult Patients With Obesity or Overweight With Weight-Related Comorbidities
Brief Title: A Study of RGT001-075 in Participants With Obesity or Overweight With Weight-Related Comorbidities
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Regor Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RGT001-075-203
Record Dates: First submitted 2024-02-01; First posted 2024-02-26 (Actual); Last update posted 2025-08-07 (Actual); Status verified 2025-08

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- RGT001-075 Group (Experimental): Patients will receive once daily dose of study drug for a total of 12 weeks
  Interventions: Drug: RGT001-075
- Placebo Group (Placebo Comparator): Patients will receive once daily dose of matching placebo for a total of 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: RGT001-075 — Administered orally
  Arms: RGT001-075 Group
Drug: Placebo — Administered orally
  Arms: Placebo Group

SUMMARY:
The main purpose of this study was to evaluate the safety and tolerability of RGT001-075 in healthy participants with obesity

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 and ≤ 75 years
* Have a BMI ≥27 kg/m² and ≤ 45 kg/m²
* Have had a stable body weight for the 3 months prior to randomization

Exclusion Criteria:

* Have obesity induced by other endocrinologic disorders or diagnosed monogenetic or syndromic forms of obesity
* Have a prior or planned surgical treatment for obesity
* Have or plan to have endoscopic and/or device-based therapy for obesity
* Have any prior diagnosis of diabetes
* Have an electrocardiogram (ECG) with abnormalities
* Have a history of Major Depressive Disorder (MDD) or other severe psychiatric disorders within the last 2 years
* Have a history of suicide attempt.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2024-03-08 (Actual); Primary Completion 2024-08-13 (Actual); Study Completion 2024-08-13 (Actual)

PRIMARY OUTCOMES:
Number of participants with Treatment-emergent Adverse Event(AE) by severity/Serious Adverse Event (SAE), with Clinical Laboratory Abnormalities, Clinically Significant Change From Baseline in Vital Signs and Abnormal Electrocardiogram(ECG) readings | 14 weeks

SECONDARY OUTCOMES:
Percent change in body weight | 12 weeks
  Percent change in body weight from baseline at Week 12
Change in body weight in kilogram | 12 weeks
  Change in body weight from baseline at Week 12
Percentage of participants who achieve ≥5% and ≥10% body weight reduction | 12 weeks
  Percentage of participants who achieve ≥5% and ≥10% body weight reduction at Week 12
Change in Body mass index (BMI) in kg/m^2 | 12 weeks
  Change in BMI from baseline at Week 12
Change in waist circumference in centimetre | 12 weeks
  Change in waist circumference from baseline at Week 12 .
RGT001-075 pharmacokinetics (PK): Area under the curve up to the last measured concentration(AUC0-last) | 12 weeks
  Analysis of AUC0-last
RGT001-075 pharmacokinetics (PK): Area under curve from time zero to time infinite(AUC0-inf) | 12 weeks
  Analysis of AUC0-inf
RGT001-075 pharmacokinetics (PK): Maximum observed concentration (Cmax) | 12 weeks
  Analysis of Cmax
RGT001-075 pharmacokinetics (PK): Time to achieve maximum concentration(Tmax) | 12 weeks
  Analysis of Tmax
RGT001-075 pharmacokinetics (PK): Elimination half-life(t1/2) | 12 weeks
  Analysis of t1/2

CONTACTS AND LOCATIONS:
Locations (10):
- United States (10):
  - Velocity Clinical Research, Los Angeles, California
  - Velocity Clinical Research, Valparaiso, Indiana
  - Velocity Clinical Research, Omaha, Nebraska
  - Velocity Clinical Research, Vestal, New York
  - Velocity Clinical Research, Durham, North Carolina
  - Velocity Clinical Research, Cleveland, Ohio
  - Velocity Clinical Research, Medford, Oregon
  - Velocity Clinical Research, East Greenwich, Rhode Island
  - Velocity Clinical Research, Dallas, Texas
  - Velocity Clinical Research, West Jordan, Utah

IPD SHARING:
Plan to Share IPD: No